CLINICAL TRIAL: NCT00583310
Title: Telephone-Based Lifestyle Intervention to Reduce Blood Pressure in Prehypertensive Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: NYU Langone Health (Other)
Collaborators: American Heart Association (Other); UNITE HERE Health Center (Unknown)
Responsible Party: Principal Investigator, Tanya Spruill, Associate Clinical Professor, Department of Medicine Behavioral Cardiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAC0714
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: High Blood Pressure
Keywords: Prehypertension
MeSH Terms: conditions — Hypertension; Prehypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Subjects receive standard written educational information at baseline, but do not receive the telephone-based intervention. Subjects may participate in the intervention following completion of the study.
- Intervention (Experimental): Four 30-minute telephone sessions including education and behavioral counseling strategies that have been shown to be effective in promoting behavior change and reducing blood pressure.
  Interventions: Behavioral: Telephone-based lifestyle counseling

INTERVENTIONS:
Behavioral: Telephone-based lifestyle counseling — Four 30-minute telephone sessions including education and behavioral counseling strategies that have been shown to be effective in promoting behavior change and reducing blood pressure.
  Arms: Intervention

SUMMARY:
Individuals with prehypertension are at risk for developing cardiovascular disease and sustained hypertension. Modifying lifestyle behaviors (diet, weight loss, sodium intake, physical activity, alcohol intake) has been shown to reduce blood pressure in hypertensives. Participants in this study will be enrolled in one of two groups. Participants in the first group will receive usual care, and participants in the second group will receive a 4 session telephone-based lifestyle intervention. The goal of the study is to determine whether this intervention is effective in promoting behavior change and reducing blood pressure among prehypertensives.

DETAILED DESCRIPTION:
Individuals with prehypertension are at increased cardiovascular risk compared with normotension, as well as increased risk of progression to sustained hypertension. The recommended treatment for prehypertension is lifestyle modification, including weight loss, adoption of the Dietary Approaches to Stop Hypertension (DASH) diet, reduction of dietary sodium, physical activity, and moderation of alcohol intake. The proposed pilot study will test the effect of a 4 session telephone-based lifestyle intervention on blood pressure change in 125 prehypertensive participants. The intervention includes education and behavioral counseling strategies that have been shown to be effective in promoting behavior change and reducing blood pressure among hypertensives.

Following baseline assessment, participants will be randomized to the intervention or usual care, and will complete follow-up assessments at 6 weeks and 3 months post-randomization. The primary aim of the study is to examine the effect of the intervention on blood pressure at 3 months. Secondary aims include examining intervention effects on lifestyle behavior changes at 6 weeks and 3 months. This study will provide pilot and feasibility data for a future application to study effects of the intervention on risk factor modification, blood pressure reduction, and cardiovascular morbidity and mortality. If successful, this brief, cost-effective intervention could easily be incorporated into routine care, and could have a significant impact on the management of prehypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Screening BP in prehypertensive range (SBP of 120-139 mmHg or DBP of 80-89 mmHg). If SBP or DBP is below these ranges, the patient is eligible. However, if either SBP or DBP is above the upper cutoffs (i.e., patient meets criteria for HTN), the patient will not be eligible.
2. Able to read and communicate in English or Spanish.
3. Must have access to a telephone at home or at work.
4. Age 18 years or older

Exclusion Criteria:

1. Patients who are currently taking anti-hypertensive medication will be excluded.
2. Patients with diabetes or kidney disease will be excluded, because pharmacologic treatment may be initiated to achieve the JNC 7 recommended BP goal of 130/80 mmHg in patients with these compelling indications.
3. Patients who are currently participating in another HTN-related clinical trial will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure change | 3 months

SECONDARY OUTCOMES:
Weight change | 3 months
Change in dietary habits | 6 weeks and 3 months
Change in physical activity level | 6 weeks and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tanya M Goyal, PhD, Principal Investigator — Columbia University; Matthew M Burg, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - UNITE HERE Health Center, New York, New York
  - Columbia University, New York, New York